CLINICAL TRIAL: NCT00357994
Title: A Randomized, Double-Blind, Double-Dummy, Efficacy, Safety and Tolerability Study of Levodopa - Carbidopa Intestinal Gel in Levodopa-Responsive Parkinson's Subjects Receiving Optimized Treatments With Parkinson Medicinal Products Who Continue to Experience Persistent Motor Fluctuations
Brief Title: Study of Efficacy, Safety and Tolerability of Levodopa-Carbidopa Intestinal Gel in Levodopa-Responsive Parkinson's Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S187.3.001; 2006-000577-29 (EudraCT Number)
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Advanced Parkinson's Disease
Keywords: carbidopa; levodopa-carbidopa; levodopa; levodopa/carbidopa suspension; dyskinesia; Duodopa; levodopa-carbidopa intestinal gel; Severe Motor Fluctuations; DUOPA
MeSH Terms: conditions — Dyskinesias | interventions — carbidopa, levodopa drug combination; Tablets; Jejunostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa-Carbidopa Intestinal Gel (LCIG) + Placebo Capsules (Experimental): Participants were randomized to LCIG (levodopa, 20 mg/mL and carbidopa monohydrate, 5 mg/mL) and placebo capsules. Participants received the percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) procedure for gel administration of LCIG.
  Interventions: Drug: Levodopa carbidopa intestinal gel (LCIG); Drug: Placebo (PBO) oral capsules; Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: PEG tube; Device: J-tube
- Placebo Gel + Levodopa-Carbidopa Capsules (Active Comparator): Participants were randomized to placebo intestinal gel and oral levodopa-carbidopa (levodopa, 100 mg and carbidopa, 25 mg) Immediate Release (IR) capsules. Participants received the percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) procedure for gel administration of placebo.
  Interventions: Drug: Placebo gel; Drug: Levodopa carbidopa (LC) oral encapsulated immediate release (IR) tablets; Device: CADD-Legacy® 1400 ambulatory infusion pump; Device: PEG tube; Device: J-tube

INTERVENTIONS:
Drug: Levodopa carbidopa intestinal gel (LCIG) — infusion should be kept within a range of 0.5-10 mL/hour (10-200 mg levodopa/hour) and is usually 2-6 mL/hour (40-120 mg levodopa per/hour)
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG) + Placebo Capsules
Drug: Placebo gel
  Arms: Placebo Gel + Levodopa-Carbidopa Capsules
Drug: Levodopa carbidopa (LC) oral encapsulated immediate release (IR) tablets
  Arms: Placebo Gel + Levodopa-Carbidopa Capsules
Drug: Placebo (PBO) oral capsules
  Arms: Levodopa-Carbidopa Intestinal Gel (LCIG) + Placebo Capsules
Device: CADD-Legacy® 1400 ambulatory infusion pump
Device: PEG tube — percutaneous endoscopic gastrostomy tube
Device: J-tube — jejunal tube

SUMMARY:
The primary objective of this study was to demonstrate the superiority of levodopa - carbidopa intestinal gel over treatment with optimized oral levodopa/carbidopa during 12 weeks.

DETAILED DESCRIPTION:
Study S187.3.001 (NCT00357994) and Study S187.3.002 (NCT00660387) were 2 identically designed, Phase 3, 12-week, randomized, double-blind, double-dummy, parallel-group, multicenter studies recruiting subjects from distinct sites. These studies evaluated the efficacy, safety, and tolerability of levodopa-carbidopa intestinal gel (LCIG) in the treatment of levodopa-responsive subjects with advanced PD who had persistent severe motor fluctuations, despite optimized treatment with oral levodopa-carbidopa, concomitant with other available antiparkinsonian medications. Participants were randomized to either LCIG active gel + placebo capsules or levodopa-carbidopa immediate release (IR) active capsules + placebo gel. Both treatment arms received the percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) procedure for gel administration, active LCIG or placebo gel. Data from these 2 studies were combined for analysis. The decision to combine the study data for analysis was made before enrollment was completed for both studies.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (PD) according to United Kingdom Parkinson's Disease Society (UKPDS) Brain Bank Criteria
* Levodopa-responsive participants who demonstrate some identifiable 'on response,' established by Investigator observation
* Demonstrate severe motor fluctuations in spite of individually optimized treatment and where therapy options are indicated

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other parkinsonian syndromes exists such as secondary parkinsonism
* Undergone surgery for the treatment of PD
* Contraindications to levodopa
* Subjects with any neurological deficit that may interfere with the study assessments

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Benesh, Study Director — AbbVie
Locations (15):
- United States (8):
  - Site Reference ID/Investigator# 45719, Los Angeles, California
  - Site Reference ID/Investigator# 45718, Englewood, Colorado
  - Site Reference ID/Investigator# 45722, Washington D.C., District of Columbia
  - Site Reference ID/Investigator# 45721, Bradenton, Florida
  - Site Reference ID/Investigator# 45705, Gainesville, Florida
  - Site Reference ID/Investigator# 45740, Baltimore, Maryland
  - Site Reference ID/Investigator# 45739, St Louis, Missouri
  - Site Reference ID/Investigator# 45703, Burlington, Vermont
- Germany (7):
  - Site Reference ID/Investigator# 44970, Bochum
  - Site Reference ID/Investigator# 44971, Bremerhaven
  - Site Reference ID/Investigator# 44973, Dresden
  - Site Reference ID/Investigator# 44965, Hanover
  - Site Reference ID/Investigator# 44964, Kiel
  - Site Reference ID/Investigator# 44966, Marburg
  - Site Reference ID/Investigator# 44968, Tübingen

REFERENCES:
- [Derived] Shih TM, Sail KR, Jalundhwala YJ, Sullivan J, van Eijndhoven E, Zadikoff C, Marshall TS, Lakdawalla DN. The effect of functional status impairment on nursing home admission risk among patients with advanced Parkinson's disease. J Med Econ. 2020 Mar;23(3):297-307. doi: 10.1080/13696998.2019.1693383. Epub 2019 Nov 28. PMID 31779508
- [Derived] Lew MF, Slevin JT, Kruger R, Martinez Castrillo JC, Chatamra K, Dubow JS, Robieson WZ, Benesh JA, Fung VS. Initiation and dose optimization for levodopa-carbidopa intestinal gel: Insights from phase 3 clinical trials. Parkinsonism Relat Disord. 2015 Jul;21(7):742-8. doi: 10.1016/j.parkreldis.2015.04.022. Epub 2015 Apr 28. PMID 25962554
- [Derived] Olanow CW, Kieburtz K, Odin P, Espay AJ, Standaert DG, Fernandez HH, Vanagunas A, Othman AA, Widnell KL, Robieson WZ, Pritchett Y, Chatamra K, Benesh J, Lenz RA, Antonini A; LCIG Horizon Study Group. Continuous intrajejunal infusion of levodopa-carbidopa intestinal gel for patients with advanced Parkinson's disease: a randomised, controlled, double-blind, double-dummy study. Lancet Neurol. 2014 Feb;13(2):141-9. doi: 10.1016/S1474-4422(13)70293-X. Epub 2013 Dec 20. PMID 24361112
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Studies S187.3.001 (NCT00357994) and S187.3.002 (NCT00660387) were 2 identically designed, Phase 3, 12-week, randomized, double-blind, double-dummy, parallel-group, multicenter studies recruiting subjects from distinct sites. All study information and results presented reflect the study data and analyses for the two studies combined.
Groups:
- LCIG + Placebo Capsules: Participants were randomized to Levodopa-Carbidopa Intestinal Gel (LCIG; levodopa, 20 mg/mL and carbidopa monohydrate, 5 mg/mL) and placebo capsules. Participants received the percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) procedure for gel administration of LCIG.
Period: Overall Study
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Started | 37 | 34
Completed | 35 | 31
Not Completed | 2 | 3
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules | Total
Number analyzed (Participants) | 37 | 34 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (9.5) | 65.1 (6.8) | 64.4 (8.3)
Age, Customized [Number; unit: participants]
  <65 years | 21 | 15 | 36
  >=65 years | 16 | 19 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Average Daily Normalized "Off" Time
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Negative change from baseline for "off" time indicates improvement.
Time Frame: Baseline, Week 12
Population: Full Analysis Set: randomized participants who had the study device implanted and had data for baseline and at least 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 31
hours | -4.04 (0.65) | -2.14 (0.66)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0015, ANCOVA — Treatment comparisons are based on an ANCOVA model including effects for treatment, country, and with the corresponding baseline and the natural logarithm of the mean daily dose of rescue medication on valid symptom diary days as covariates; Treatment Difference (LS Mean) = -1.91, 95% CI 2-sided [-3.05 to -0.76], Standard Error of Mean 0.57

2. Secondary Outcome: Change From Baseline in Average Daily Normalized "On" Time Without Troublesome Dyskinesia at Week 12
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. "On" time without troublesome dyskinesia (involuntary muscle movement) is defined as "on" time without dyskinesia and "on" time with non-troublesome dyskinesia. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis. Positive change from Baseline for "on" time without troublesome dyskinesia indicates improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: hours
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 31
hours | 4.11 (0.75) | 2.24 (0.76)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Since the null hypothesis for the primary analysis was rejected in favor of the alternative hypothesis, hierarchical testing was performed for secondary variables on the Full Analysis data set at the 0.50 level using a gatekeeping procedure to preserve family-wise error rate; Test type: Superiority or Other; p = 0.0059, ANCOVA; Treatment comparisons are based on an ANCOVA model including effects for treatment, country, and with the corresponding baseline as a covariate; Treatment Difference (LS Mean) = 1.86, 95% CI 2-sided [0.56 to 3.17], Standard Error of Mean 0.65

3. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Summary Index at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. These include: mobility, activities of daily living, emotional well-being, stigma, social support, cognition, communication, and bodily discomfort. The PDQ-39 Summary Index is the sum of all answers divided by the highest score possible (i.e. number of answers multiplied by 4) which is multiplied by 100 to put the score on a 0-100 scale. Higher scores are associated with more severe symptoms.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -10.9 (3.3) | -3.9 (3.2)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0155, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -7.0, 95% CI 2-sided [-12.6 to -1.4], Standard Error of Mean 2.8

4. Secondary Outcome: Clinical Global Impression - Status (CGI-S) Score at Baseline and Clinical Global Impression - Improvement (CGI-I) Score at Week 12
Description: The CGI-S is a global assessment by the Investigator of current symptomatology and impact of illness on functioning. The ratings of the CGI-S are as follows: 1 = normal, 2 = borderline ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, and 7 = among the most extremely ill. The CGI-I is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-I ratings are as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, 7 = very much worse.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale
  CGI-S at Baseline | 4.2 (0.7) | 4.6 (0.8)
  CGI-I at Week 12 | 2.3 (1.2) | 3.2 (1.4)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0258, ANCOVA; Treatment comparisons are based on an ANCOVA model including effects for treatment, country, and with the baseline CGI-S as a covariate; Treatment Difference (LS Mean) = -0.7, 95% CI 2-sided [-1.4 to -0.1], Standard Error of Mean 0.3

5. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part II Score at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions that comprise Part II, each of which are measured on a 5-point scale (0-4). The Part II score ranges from 0-52 and higher scores are associated with more disability.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -1.8 (1.3) | 1.3 (1.3)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0086, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -3.0, 95% CI 2-sided [-5.3 to -0.8], Standard Error of Mean 1.1

6. Secondary Outcome: Change From Baseline in UPDRS Part III Score at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part III score is the sum of the 27 answers provided to the 14 Part III questions, each of which are measured on a 5-point scale (0-4). The Part III score ranges from 0-108 and higher scores are associated with more disability.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -1.5 (2.4) | -2.9 (2.4)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.5020, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = 1.4, 95% CI 2-sided [-2.8 to 5.6], Standard Error of Mean 2.1

7. Secondary Outcome: Change From Baseline in EuroQual Quality of Life - 5 Dimensions (EQ-5D) Summary Index at Week 12
Description: The EQ-5D is a participant answered questionnaire scoring 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ-5D health states, defined by the EQ-5D descriptive system, are converted into a single summary index by applying a formula that essentially attaches values (also called QOL weights or QOL utilities) to each of the levels in each dimension. EQ-5D Summary Index values range from -0.11 to 1.00 with positive change indicating improvement.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 32
units on a scale | 0.054 (0.043) | -0.016 (0.043)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0670, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = 0.070, 95% CI 2-sided [-0.005 to 0.146], Standard Error of Mean 0.038

8. Secondary Outcome: Change From Baseline in Zarit Burden Interview (ZBI) Total Score at Week 12
Description: The ZBI is a 22-item questionnaire regarding the caregiver/subject relationship and evaluates the caregiver's health condition, psychological well-being, finances and social life. Each question is answered on a 5-point scale (0=Never, 1=Rarely, 2=Sometimes, 3=Quite frequently, and 4= Nearly always). The caregiver burden is evaluated by the total score (Range 0 to 88) obtained from the sum of the answers to the 22 questions. Higher scores are associated with a higher level of burden for the caregiver.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 23 | 23
units on a scale | -2.8 (3.7) | 1.7 (3.3)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1501, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treament Difference (LS Mean) = -4.5, 95% CI 2-sided [-10.7 to 1.7], Standard Error of Mean 3.1

9. Secondary Outcome: Change From Baseline in Average Daily Normalized "On" Time With Troublesome Dyskinesia at Week 12
Description: Based on the Parkinson's Disease Symptom Diary. "On" time is when PD symptoms are well controlled by the drug. "Off" time is when PD symptoms are not adequately controlled by the drug. The diary is completed every 30 minutes for the full 24 hours of each of 3 days prior to selected clinic visits. It reflects both time awake and time asleep. Daily totals are normalized to a 16-hour scale (i.e. 16 hours of awake time). The normalized totals for the 3 days prior to the visit are averaged for the analysis.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 31
units on a scale | -0.11 (0.52) | -0.03 (0.52)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.8574, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -0.08, 95% CI 2-sided [-0.98 to 0.82], Standard Error of Mean 0.45

10. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Mobility Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Mobility (e.g., fear of falling when walking) includes 10 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -17.3 (5.0) | -6.8 (4.9)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0184, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -10.4, 95% CI 2-sided [-19.1 to -1.8], Standard Error of Mean 4.3

11. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Activities of Daily Living Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Activities of Daily Living (e.g., difficulty cutting food) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -12.9 (5.3) | -1.3 (5.2)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0129, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -11.6, 95% CI 2-sided [-20.6 to -2.5], Standard Error of Mean 4.5

12. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Emotional Well-Being Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Emotional Well-being (e.g., feelings of isolation) includes 6 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 32
units on a scale | -7.1 (4.0) | -4.9 (4.0)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.5246, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -2.2, 95% CI 2-sided [-9.0 to 4.6], Standard Error of Mean 3.4

13. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Stigma Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Stigma (e.g., social embarrassment) consists of 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -8.9 (4.4) | -4.5 (4.4)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.2423, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -4.5, 95% CI 2-sided [-12.0 to 3.1], Standard Error of Mean 3.8

14. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Social Support Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Social Support includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 32
units on a scale | -3.9 (3.5) | -0.1 (3.6)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.2243, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -3.8, 95% CI 2-sided [-9.9 to 2.4], Standard Error of Mean 3.1

15. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Cognition Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Cognition includes 4 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -7.3 (4.0) | -3.2 (3.9)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.2407, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -4.0, 95% CI 2-sided [-10.8 to 2.8], Standard Error of Mean 3.4

16. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Communication Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Communication includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -9.5 (4.1) | 4.4 (4.1)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -13.8, 95% CI 2-sided [-20.8 to -6.8], Standard Error of Mean 3.5

17. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39) Bodily Discomfort Domain Score at Week 12
Description: The PDQ-39 is a self-administered questionnaire which comprises 39 items addressing 8 domains of health in Parkinson's disease patients. The PDQ-39 Domain: Bodily Discomfort includes 3 questions, each answered on a 5-point scale. The domain scores are calculated by first summing the answers to the questions in the domain. The sum is divided by the highest score possible (i.e., number of answers multiplied by 4) and the quotient is multiplied by 100 to put the score on a scale from 0 to 100, where lower scores indicate a better perceived health status. Higher scores are consistently associated with the more severe symptoms of the disease such as tremor and stiffness.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -13.5 (6.1) | -10.2 (6.0)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.5213, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -3.3, 95% CI 2-sided [-13.6 to 6.9], Standard Error of Mean 5.1

18. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part I Score at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part I Score is the sum of the answers to the 4 questions that comprise Part I, each of which are measured on a 5-point scale (0-4). The Part I score ranges from 0-16 and higher scores are associated with more disability.
Time Frame: Baseline, Week 12
Population: Full Analysis Set: randomized participants who had the study device implanted and had data for baseline and at least 1 post-baseline assessment. No missing data was imputed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -0.2 (0.4) | -0.5 (0.4)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.3741, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = 0.3, 95% CI 2-sided [-0.4 to 0.9], Standard Error of Mean 0.3

19. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Score at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part IV Score is the sum of the answers to the 11 questions that comprise Part IV, each of which are measured on a 5-point scale (0-4) or a 2-point scale (0 or 1). The Part IV score ranges from 0-23 and higher scores are associated with more disability.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -1.1 (0.7) | 0.1 (0.7)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0361, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -1.2, 95% CI 2-sided [-2.4 to -0.1], Standard Error of Mean 0.6

20. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part IV Questions 32, 33, and 34 at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. Questions 32, 33, and 34 on UPDRS Part IV were totaled to evaluate dyskinesias. Each of these questions is measured on a 5-point scale (0-4). The Part IV dyskinesia score will range from 0-12 and higher scores are associated with more disability.
Time Frame: Baseline, Week 12
Population: as for outcome 18
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | 0.4 (0.5) | 0.8 (0.5)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.3578, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -0.4, 95% CI 2-sided [-1.1 to 0.4], Standard Error of Mean 0.4

21. Secondary Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Total Score at Week 12
Description: The UPDRS is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The total score is the sum of the responses to the 31 questions (44 answers) that comprise Parts I-III of the scale. The total score will range from 0-176, with 176 representing the worst (total) disability, and 0 no disability.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 33
units on a scale | -3.6 (3.4) | -2.1 (3.4)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.6088, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = -1.5, 95% CI 2-sided [-7.4 to 4.4], Standard Error of Mean 2.9

22. Secondary Outcome: Change From Baseline in EuroQol Quality of Life Scale (EQ-5D) Visual Analogue Scale (VAS) at Week 12
Description: The EQ-5D VAS records the participant's self-rated health on a scale from 0-100 where 100 is the 'best imaginable health state' and 0 is the 'worst imaginable health state.'
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 36 | 32
units on a scale | 5.2 (4.3) | -6.3 (4.3)
Statistical Analysis 1: Comparison: LCIG + Placebo Capsules vs Placebo Gel + Levodopa-Carbidopa Capsules; Test type: Superiority or Other; p = 0.0033, ANCOVA; [statistical method as in outcome 2, analysis 1]; Treatment Difference (LS Mean) = 11.4, 95% CI 2-sided [4.0 to 18.9], Standard Error of Mean 3.7

23. Secondary Outcome: Employment Impairment (EMP) I Status at Baseline
Description: The EMP instruments are designed to collect information regarding employment and ability to run a household. EMP I questions include: Are you currently in paid employment? (If yes, at which percentage have you been working during the last 4 weeks?); Have you got someone to run your household for you? (If yes, how much time per week does he/she spend in your household?); Are you retired? (If yes, for which reason?).
Time Frame: Baseline
Population: Full Analysis Set: randomized participants who had the study device implanted and had data for baseline and at least 1 post-baseline assessment. Missing data was not imputed.
Measure: Number; unit: participants
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 31
participants
  Paid Employment (PE)=Yes | 10 | 8
  PE=Yes, 100% of Past 4 Weeks | 6 | 3
  PE=Yes, 75% of Past 4 Weeks | 2 | 1
  PE=Yes, 50% of Past 4 Weeks | 0 | 2
  PE=Yes, 25% of Past 4 Weeks | 1 | 1
  PE=Yes, Other % of Past 4 Weeks | 1 | 1
  PE=No | 25 | 23
  Someone Else Runs the Household (SRH)=Yes | 24 | 25
  SRH=Yes, 100% of Time per Week | 15 | 13
  SRH=Yes, 75% of Time per Week | 3 | 4
  SRH=Yes, 50% of Time per Week | 3 | 5
  SRH=Yes, 25% of Time per Week | 2 | 1
  SRH=Yes, Other % of Time per Week | 1 | 2
  SRH=No | 11 | 6
  Are You Retired (R)=Yes | 24 | 23
  R=Yes, Old Age Pensioner | 8 | 8
  R=Yes, Premature Due to PD | 13 | 12
  R=Yes, Premature Due to Other Condition | 1 | 1
  R=Yes, Other Reason | 2 | 2
  R=No | 11 | 8

24. Secondary Outcome: Employment Impairment (EMP) II Status at Week 12
Description: The EMP instruments are designed to collect information regarding employment and ability to run a household. EMP I questions include: Are you currently in paid employment? (If yes, at which percentage have you been working during the last 4 weeks?); Have you got someone to run your household for you? (If yes, how much time per week does he/she spend in your household?); Are you retired? (If yes, for which reason?) The retirement question (from EMP I) is excluded from the EMP II instrument.
Time Frame: Week 12 (or early termination)
Population: as for outcome 23
Measure: Number; unit: participants
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Number analyzed (Participants) | 35 | 31
participants
  Paid Employment (PE)=Yes | 10 | 5
  PE=Yes, 100% of Past 4 Weeks | 6 | 1
  PE=Yes, 75% of Past 4 Weeks | 1 | 1
  PE=Yes, 50% of Past 4 Weeks | 1 | 2
  PE=Yes, 25% of Past 4 Weeks | 0 | 1
  PE=Yes, Other % of Past 4 Weeks | 2 | 0
  PE=No | 25 | 26
  Someone Else Runs the Household (SRH)=Yes | 22 | 24
  SRH=Yes, 100% of Time per Week | 13 | 12
  SRH=Yes, 75% of Time per Week | 5 | 4
  SRH=Yes, 50% of Time per Week | 0 | 4
  SRH=Yes, 25% of Time per Week | 2 | 2
  SRH=Yes, Other % of Time per Week | 2 | 2
  SRH=No | 13 | 7

ADVERSE EVENTS:
Time Frame: From Screening to the end of study or early termination of treatment, including the removal of PEG-J (up to 12 weeks), plus 30 days.
Description: Serious adverse events (AEs) and treatment-emergent AEs are presented. Treatment-emergent adverse events were defined as AEs that began or worsened from date of the study device implantation to the end of therapy (last dose of study drug or PEG-J removal, whichever is later) plus 30 days.
Groups:
- LCIG + Placebo Capsules: Participants were randomized to Levodopa-Carbidopa Intestinal Gel (LCIG; levodopa, 20 mg/mL and carbidopa, 5 mg/mL) and placebo capsules. Participants received the percutaneous endoscopic gastrostomy with jejunal extension (PEG-J) procedure for gel administration of LCIG.
Arm/Group | LCIG + Placebo Capsules | Placebo Gel + Levodopa-Carbidopa Capsules
Serious Adverse Events (participants affected / at risk) | 5/37 | 7/34
Other Adverse Events (participants affected / at risk) | 35/37 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCIG + Placebo Capsules (N=37) | Placebo Gel + Levodopa-Carbidopa Capsules (N=34)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 0 | 1
PNEUMOPERITONEUM (Gastrointestinal disorders) | 1 | 0
COMPLICATION OF DEVICE INSERTION (General disorders) | 1 | 1
CATHETER SITE CELLULITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 2
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
BODY TEMPERATURE INCREASED (Investigations) | 0 | 1
SPINAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 0 | 1
DYSKINESIA (Nervous system disorders) | 1 | 0
HYPERSOMNIA (Nervous system disorders) | 1 | 0
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0
DELUSION (Psychiatric disorders) | 1 | 0
HALLUCINATION (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1
MUTISM (Psychiatric disorders) | 1 | 0
PSYCHOTIC DISORDER (Psychiatric disorders) | 1 | 1
RENAL CYST (Renal and urinary disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCIG + Placebo Capsules (N=37) | Placebo Gel + Levodopa-Carbidopa Capsules (N=34)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 | 3
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 19 | 10
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 2
CONSTIPATION (Gastrointestinal disorders) | 8 | 7
DIARRHOEA (Gastrointestinal disorders) | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 2 | 1
FLATULENCE (Gastrointestinal disorders) | 6 | 4
GASTRITIS (Gastrointestinal disorders) | 1 | 3
HIATUS HERNIA (Gastrointestinal disorders) | 3 | 2
NAUSEA (Gastrointestinal disorders) | 11 | 7
PNEUMOPERITONEUM (Gastrointestinal disorders) | 3 | 1
REFLUX OESOPHAGITIS (Gastrointestinal disorders) | 0 | 2
VOMITING (Gastrointestinal disorders) | 2 | 4
COMPLICATION OF DEVICE INSERTION (General disorders) | 20 | 14
FATIGUE (General disorders) | 0 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 2
OEDEMA PERIPHERAL (General disorders) | 3 | 0
PYREXIA (General disorders) | 2 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 4 | 8
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 4
FALL (Injury, poisoning and procedural complications) | 4 | 4
INCISION SITE ERYTHEMA (Injury, poisoning and procedural complications) | 7 | 4
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 4 | 3
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 2 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 11 | 12
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 2 | 2
BACTERIAL TEST POSITIVE (Investigations) | 2 | 0
VITAMIN B6 DECREASED (Investigations) | 1 | 2
WEIGHT DECREASED (Investigations) | 0 | 2
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 2 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 5
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 2
DIZZINESS (Nervous system disorders) | 3 | 2
DYSKINESIA (Nervous system disorders) | 4 | 4
FREEZING PHENOMENON (Nervous system disorders) | 1 | 2
HEADACHE (Nervous system disorders) | 3 | 4
ANXIETY (Psychiatric disorders) | 3 | 1
DEPRESSION (Psychiatric disorders) | 4 | 1
INSOMNIA (Psychiatric disorders) | 4 | 4
SLEEP DISORDER (Psychiatric disorders) | 2 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 3 | 0
EXCESSIVE GRANULATION TISSUE (Skin and subcutaneous tissue disorders) | 2 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 3 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.